CLINICAL TRIAL: NCT01554813
Title: A Single - Blind, Randomized, - Controlled Clinical Trial With Inactivated Influenza Vaccine (Split Virion) (0.5ml Formulation)
Brief Title: Clinical Trial of Inactivated Influenza Vaccine (0.5ml Formulation)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hualan Biological Engineering, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Hualanbio-influenza III-001; Hualanbio-phase III-001 (Other Grant/Funding Number: Hualan Biological Engineering Inc.)
Record Dates: First submitted 2012-03-12; First posted 2012-03-15 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-03

CONDITIONS: Influenza
Keywords: Influenza Vaccine, Vaccination,
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Influenza split vaccine of 15μg HA (Experimental): 15μg HA/strain/0.5ml/vial
  Interventions: Biological: Influenza split vaccine of 15 μg HA
- Influenza split vaccine of 15 μg HA (Experimental): 15μg HA/strain/0.5ml/syringe
  Interventions: Biological: Influenza split vaccine of 15 μg HA
- Influenza split vaccine (Active Comparator): 15μg HA/strain/0.5ml/syringe
  Interventions: Biological: Influenza split vaccine

INTERVENTIONS:
Biological: Influenza split vaccine of 15 μg HA — 60 subjects were assigned (20 infants, 20 children and 20 adults) to receive influenza vaccine (split virion), inactivated, 0.5ml, one dose regime
  Other Names: Hualan Bio
  Arms: Influenza split vaccine of 15 μg HA; Influenza split vaccine of 15μg HA
Biological: Influenza split vaccine of 15 μg HA — 558 subjects were assigned to receive influenza split vaccine, 0.5ml, one dose regime
  Other Names: Hualan Bio
  Arms: Influenza split vaccine of 15 μg HA; Influenza split vaccine of 15μg HA
Biological: Influenza split vaccine — 280 subjects were assigned to receive influenza split vaccine, 0.5ml, one dose regime
  Other Names: Shenzhen Aventis Pasteur
  Arms: Influenza split vaccine

SUMMARY:
The clinical trial was conducted in Jintan City of Jiangsu Province, China in May, 2006. The purpose of the clinical trial was to evaluate the safety and immunogenicity against Hualan's Influenza Vaccine (Split Virion), Inactivated (0.5ml) administered on age 6 months and old population.

DETAILED DESCRIPTION:
The clinical trial was designed randomized and blind. Participants included up to 900 persons. The clinical trial had two stages: the first stage selected 60 subjects to be administered test vaccine for preliminary safety study; 840 subjects were selected at the second stage for the observation of the safety and immunogenicity against the test vaccine administered on large population on the basis of the first stage. There were 560 subjects and 280 subjects in the test group and control group respectively.

Venous blood from subjects was collected before immunization and 4 weeks after the whole immunization for the analysis of the immunogenicity. The information about adverse reactions/time was reported to the SFDA every month during the trial under the status of blinding. Unblinding was conducted after the subject follow-up and observation.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria for the primary vaccination on subjects over 3 years old and subjects 6 months～3 years old

   * Healthy male and female 6 months or over, subject (or their guardians) are able to understand and sign informed consent
   * Healthy person by inquiring illness history, physical examination and clinical judgment and who complies with vaccination of this product
   * Be able to comply with the requirement of clinical trial protocol
   * Have no history of influenza vaccination within the past 6 months and vaccination with other product within the latest 1 week;
   * Axillary temperature<37.1℃.
2. Inclusion criteria for the boost vaccination on subjects age 6 months～3 years

   * Have no history of vaccination with other preventive product within the latest 1 week;
   * Axillary temperature<37.1℃.

Exclusion Criteria:

1. Exclusion criteria for the primary vaccination on subjects over 3 years old and subjects age 6 months～3 years

   * Serious diseases, such as: tumor, autoimmunity disease, progressive atherosclerotic disease or diabetes with complication, COPD needing oxygen uptake treatment, acute or progressive liver or kidney disease, CHF, etc.
   * Subjects who are allergic to any component of test vaccine (history of vaccination allergy), especially allergic to eggs
   * History of symptoms or signs in neurological system
   * Known or suspected (high risk of onset) damaged or abnormal immunologic function need receiving immunosuppressant or immunopotentiator treatment; history of receiving immunoglobulin or blood product or plasma extractive outside the gastrointestinal tract within the past 3 months; and HIV infection or relevant diseases
   * Haemorrhage physique or extension of haemorrhage time
   * History of influenza or at least once influenza vaccination within the past 6 months
   * History of receiving other vaccination or injection of immunoglobulin and any test drug within the past 1 week
   * History of any acute disease and infection needing antibiotics or antiviral treatment in whole body within the past 7 days
   * History of fever within the past three days (axillary temperature≥37.1℃)
   * Participating in another clinical trial
   * History of allergy, eclampsia, epilepsy, encephalopathy and mental disease or family disease;
   * Thrombopenia or other coagulopathy that may cause contraindication of intramuscular injection
   * Serious chronic disease (such as Down syndrome, diabetes, sickle cell anemia or neurologic disease, and GBS)
   * Known or suspected diseases at the same time, including: respiratory system disease, acute infection or active stage of chronic disease, HIV infection of infants or mothers, CVD, serious hypertension, during the treatment of tumor and skin disease
   * Any condition may affect trial assessment in judgment of investigators.
2. Exclusion criteria for the boost vaccination on subjects age 6 months～3 years

   * History of receiving other vaccination or injection of immunoglobulin and any test drug within the past 1 week
   * History of any acute disease and infection needing antibiotics or antiviral treatment in whole body within the past 7 days
   * History of fever within the past three days (axillary temperature≥37.1℃).

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2006-05; Primary Completion 2006-07 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety study | 28 days after the vaccination
  Include ADR, adverse event and severe adverse event.

SECONDARY OUTCOMES:
Observation of immunogenicity | 28 days after the immunization
  The rate of seroconversion, the rate of seroprotection, the GMT, and the antibody increasing folds of the subjects after administration with the vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Feng-cai Zhu, M.D., Study Director — Jiangsu Provicial Center for Disease Provention and Control
Locations (1):
- Jiangsu Provincial Center for Disease Prevention and Control, Nanjing, Jiangsu, China